CLINICAL TRIAL: NCT06544096
Title: Evaluation of the Effectiveness of a Neonatal Home Skin Care Guidance Based on We-chat: A Cluster-Randomized Controlled Trial
Brief Title: Application Evaluation of Newborn Home Skin Care Management System Under the Service of "WeChat Platform+Health Care"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024/6/7
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Infants
MeSH Terms: interventions — Delivery of Health Care; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (Active Comparator): Routine health education
  Interventions: Behavioral: control group (routine health education)
- Using"WeChat platform+health care" group (Experimental): Use"WeChat platform+health care"
  Interventions: Behavioral: intervention group (WeChat platform + healthcare)

INTERVENTIONS:
Behavioral: intervention group (WeChat platform + healthcare) — The study will implement the WeChat-based Neonatal Home Skin Care Management System, designed based on neonatal skin characteristics and evidence-based care guidelines. The intervention materials included a WeChat platform functional module (comprising a newborn information registration interface, online consultation, and questionnaire features) along with standard educational brochures used in the control group. During hospitalization, study group healthcare providers will deliver standard health education (identical to the control group) while additionally guiding mothers through platform registration and data entry, with demonstrations of system functionality. Post-discharge, the system automatically will deliver stage-appropriate skin care recommendations based on neonatal age with read reminders prompting parental engagement. Parents can access educational materials or submit queries at any time, while researchers utilize the platform for survey distribution.
  Arms: Using"WeChat platform+health care" group
Behavioral: control group (routine health education) — When the parturient is discharged from the hospital, the medical staff of the control unit will give the parturient health education about the discharge of the newborn. The contents of the education include neonatal jaundice, umbilical care, vaccination, 42-day follow-up, breastfeeding and so on, which are not included in the system.
  Arms: the control group

SUMMARY:
Through the establishment of the newborn home skin care management system under the service of "WeChat platform+health care", the investigators focus on the common skin problems of newborns at home, push health education materials through the system, teach parents the methods and details of home skin care, and evaluate the effect of the system on reducing the incidence of newborn home skin problems and the prognosis of home skin problems through cluster randomized controlled research.

DETAILED DESCRIPTION:
In this study, the cluster randomization method is used, and eight centers are assigned to the experimental group or the control group according to the ratio of 1:1. Randomization plan is made by independent statistical team in statistical software: by creating random seed numbers and sorting them, the intervention plan distribution of each center is determined. The outcome evaluator and the statistical analysis team will not know the grouping situation of each center.

In this study, there are 4 centers in the experimental group and 4 centers in the control group. Sample size calculation is based on the main outcome index: the incidence of diaper dermatitis in newborns at home.

ELIGIBILITY:
Inclusion Criteria:

* Newborns born in normal delivery (gestational age ≧35w)
* Newborns' parents can cooperate, have certain learning, reading and understanding abilities, and have the ability to care for newborns
* Voluntary participation in this study.

Exclusion Criteria:

* Newborns requiring hospitalization.
* Newborns diagnosed with congenital skin diseases.
* The newborn mother has mental illness.
* The newborn mother has a serious illness and needs hospitalization.

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 692 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of diaper dermatitis in newborns at home | Within two months after birth
  The proportion of people with diaper dermatitis in the total number of people in the study.The diagnosis of diaper dermatitis is based on any rash in the diaper area reported by parents.

SECONDARY OUTCOMES:
Incidence rate of neonatal home atopic dermatitis (AD) | Within two months after birth
  The proportion of people with atopic dermatitis (AD) in the total number of people in the study.The subjects reported by parents are itching, typical morphology and location (flexor dermatitis) or atypical morphology and location accompanied by xeroderma and chronic or recurrent course of disease; Have the above three items at the same time to diagnose.
Rate of Hospital Visits for Skin Problems | Within two months after birth
  The rate of parent-initiated hospital visits for infant skin problems was calculated as the total number of visits for skin issues divided by the total number of newborns investigated during the study period.
Parental Knowledge of Home Skincare | Within two months after birth
  Parental knowledge of home skincare was assessed using questionnaire scores on skin management knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Hu Xiaojing, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang T, Chen Y, Dou Y, Qiu M, Wang Y, Jiang S, Hu X. Parent-guided home skin care for infants via a WeChat platform: a study protocol for a cluster randomized controlled trial. Trials. 2025 Oct 31;26(1):458. doi: 10.1186/s13063-025-09186-x. PMID 41174684